CLINICAL TRIAL: NCT03085160
Title: Project EAT: Eating and Attitudes in Teens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 14-5084
Record Dates: First submitted 2017-03-09; First posted 2017-03-21 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Obesity; Adolescent Development; Stress
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Learning to Breathe (Experimental): Six-week mindfulness-based group program for adolescents
  Interventions: Behavioral: Learning to Breathe
- Health Education (Active Comparator): Six-week health education group program for adolescents
  Interventions: Behavioral: Health Education

INTERVENTIONS:
Behavioral: Learning to Breathe — Six-session group program that involves meditation and interactive activities to learn mindfulness skills for coping with stress
  Arms: Learning to Breathe
Behavioral: Health Education — Six-session group program that covers topics important for healthy living such as avoiding drug use, conflict resolution, bullying, sun safety and others
  Arms: Health Education

SUMMARY:
Research suggests there is a connection between mood and weight. People who feel stressed or depressed are more likely to be overweight than people who don't have these feelings. Some individuals turn to food to cope, which can lead to gaining too much weight over time. Adolescence is an important time to understand these connections. Patterns of handling stress learned during adolescence set the stage for stress management in adulthood. This study is a randomized controlled pilot study with 60 adolescents who are at-risk for future, chronic obesity. The investigators will test if taking part in a 6-week group program to lower stress and improve mood will be helpful to teens at-risk.

ELIGIBILITY:
Inclusion Criteria:

* Age 12-17 years
* At-risk for long-term obesity by virtue of current BMI (≥70th percentile for age and sex) or obesity (BMI ≥30 kg/m2) in both biological parents
* Good general health

Exclusion Criteria:

* Current full-syndrome psychiatric disorder that in the investigators' opinion would impede study compliance
* Major medical problem such as type 2 diabetes
* Use of medication affecting mood or body weight such as stimulants or anti-depressants
* Any medical issues that could be acutely worsened by exercise such as asthma or musculoskeletal problems.
* Pregnancy in females

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2014-10-27 (Actual); Primary Completion 2020-12-05 (Actual); Study Completion 2020-12-05 (Actual)

PRIMARY OUTCOMES:
Feasibility of study | 3 years
  Rate of recruitment of eligible adolescent volunteers
Acceptability of program | 6 weeks
  Session attendance determined as percentage of total sessions (6) attended
Acceptability of study participation | 6 weeks
  Post-intervention acceptability ratings

SECONDARY OUTCOMES:
Perceived stress | 6 months
  Changes in perceived stress as assessed by the 10-item version Perceived Stress Scale total score, computed as the sum of all items (range 0-40) with higher scores indicating greater perceived stress
Executive function | 6 months
  Executive function assessed with the parent version of the Behavior Rating Inventory of Everyday Executive Function, with 8 subscales computed as the sum of their respected items, including inhibit (range 0-20), shift (range 0-16), emotional control (range 0-20), initiate (range 0-16), working memory (range 0-20), planning/organization (range 0-24), organization of materials (range 0-12), and monitor (range 0-16). Higher scores reflect more problematic executive dysfunction
Food reward sensitivity | 6 months
  Relative reinforcing value of food assessed with behavioral task, with the outcome being the shift point when individuals shift from choosing a palatable food reward to an alternative reward (range 20-240) with higher scores reflecting greater sensitivity to food as a reward
Meal intake | 6 months
  Measured laboratory test meal intake
Weight gain | 6 months
  Gain in BMI (kg/m2) units
Fat gain | 6 months
  Gain in body fat mass as measured by air displacement plethysmography

CONTACTS AND LOCATIONS:
Locations (1):
- Colorado State University, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shomaker LB, Berman Z, Burke M, Annameier SK, Pivarunas B, Sanchez N, Smith AD, Hendrich S, Riggs NR, Legget KT, Cornier MA, Melby C, Johnson SA, Lucas-Thompson R. Mindfulness-based group intervention in adolescents at-risk for excess weight gain: A randomized controlled pilot study. Appetite. 2019 Sep 1;140:213-222. doi: 10.1016/j.appet.2019.05.022. Epub 2019 May 18. PMID 31112737